CLINICAL TRIAL: NCT02041871
Title: Interest of Preoperative Immunonutrition in Liver Resection for Cancer
Brief Title: Interest of PReOPerative Immunonutrition in Liver Surgery for Cancer
Acronym: PROPILS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Nestlé Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P120207
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-02

CONDITIONS: Hepatectomy; Elective Hepatectomy; Malignant Tumors
Keywords: Liver Surgery; Hepatectomy; Immunonutrition; Cancer; Morbidity; Postoperative complication
MeSH Terms: conditions — Neoplasms; Postoperative Complications | interventions — Immunonutrition Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Impact control (Experimental): ORAL IMPACT Powder 74g within 250ml of water, 3 times per day during 7 days before surgery
  Interventions: Dietary Supplement: Oral immunonutrition
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oral immunonutrition — Powder 74g within 250ml of water, 3 times per day during 7 days before surgery
  Other Names: ORAL IMPACT
  Arms: Impact control
Dietary Supplement: Placebo — Powder 74g within 250ml of water, 3 times per day during 7 days before surgery
  Arms: Placebo

SUMMARY:
To study the efficacy of preoperative immunonutrition in reducing postoperative morbidity after liver resection for cancer.

DETAILED DESCRIPTION:
Perioperative immunonutrition has been developed to improve the immuno metabolic host response and outcome in postoperative period and has been proven to be beneficial in reducing significantly postoperative infectious complications and length of hospital stay in patients undergoing elective gastrointestinal surgery for tumors. To date, the effects of preoperative oral immunonutrition (ORAL IMPACT) in non cirrhotic patients undergoing liver resection for cancer are unknown. The purpose of this study is to determine whether the administration of a short-term preoperative oral immunonutrition can reduce postoperative morbidity in non-cirrhotic patients undergoing liver resection for malignant tumours.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Non cirrhotic patient
* Elective liver surgery for cancer (primary or secondary malignant tumours)
* Hepatectomy including at least 1 segment or 3 wedge resections

Exclusion Criteria:

* Liver resection for benign lesions
* Liver resection associated with biliary tract surgery
* Liver resection associated with gastro-intestinal surgery
* Cirrhosis, defined by transient elastography (Fibroscan®) or by liver biopsy
* Renal failure
* Pregnancy or nursing women
* History of hypersensitivity or allergy to arginine, omega-3 fatty acids, or nucleotides
* Inability to take oral nutrition
* Mental condition rendering the subject unable to understand the nature, end-points and consequences of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2013-09; Primary Completion 2018-09-13 (Actual); Study Completion 2018-09-13 (Actual)

PRIMARY OUTCOMES:
Overall complications classified in grade 2-3-4 or 5 by DINDO-CLAVIEN | In the first 30 postoperative days after Liver surgery

SECONDARY OUTCOMES:
Length of hospital stay | 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Denis CASTAING, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP, Paul Brousse Hospital, Centre Hepato-Biliaire, Villejuif, France

REFERENCES:
- [Derived] Ciacio O, Voron T, Pittau G, Lewin M, Vibert E, Adam R, Sa Cunha A, Cherqui D, Schielke A, Soubrane O, Scatton O, Salloum C, Azoulay D, Benoist S, Goyer P, Vaillant JC, Hannoun L, Boleslawski E, Agostini H, Samuel D, Castaing D. Interest of preoperative immunonutrition in liver resection for cancer: study protocol of the PROPILS trial, a multicenter randomized controlled phase IV trial. BMC Cancer. 2014 Dec 18;14:980. doi: 10.1186/1471-2407-14-980. PMID 25523036